CLINICAL TRIAL: NCT05527132
Title: Understanding the Phenomena of Aging and Rupture of Breast Implants
Acronym: CRIMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8528
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Aging of Breast Implants
Keywords: Breast Prosthesis Implantation; Aging of breast implants; Rupture of breast implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast implants, like all implantable medical devices, are subject to wear and tear as they age in the body. In addition to this wear and tear, they are subject to external trauma, whether accidental during daily life, during insertion or during mammography.

The kinetics and mechanisms of aging are poorly studied and the phenomenon of implant rupture is not elucidated. However, studies of older generation implants have shown that implant rupture is correlated with the duration of implantation.

ELIGIBILITY:
Inclusion criteria:

* Female adult (≥18 years old)
* operated on at the HUS for a change of breast prosthesis, aesthetic or reconstruction, between 2022 and 2024
* having not expressed, after information, her opposition to participate in this research.

Exclusion criteria:

* Women who have expressed their opposition to participating in the study
* ruptured prosthesis, associated with a LAGC-AIM, excessive perspiration
* interfering treatments and associated diseases, history

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Female adult (≥18 years old) operated on at the HUS for a change of breast prosthesis, aesthetic or reconstruction, between 2022 and 2024
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
The mechanical properties of breast implants will be evaluated by uniaxial tensile tests | After extraction of breast implants

CONTACTS AND LOCATIONS:
Overall Officials: laetitia RUFFENACH, MD, Principal Investigator — Service de Chirurgie Plastique Esthétique et Reconstructrice - CHU de Strasbourg - France
Locations (1):
- Service de Chirurgie Plastique Esthétique et Reconstructrice - CHU de Strasbourg - France, Strasbourg, France